CLINICAL TRIAL: NCT05014529
Title: The Continuous Positive Airway Pressure Effect on Rho-associated Coiled-coil Containing Kinases Activity and Left Ventricle Mass in Obstructive Sleep Apnea-hypopnea Syndrome.
Brief Title: The Continuous Positive Airway Pressure Effect on Rho-associated Coiled-coil Containing Kinases Activity.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chung-Chieh, Yu, Director of Pulmonary Medicine Division, Chang Gung Memorial Hospital
Other Study IDs: 202009223870
Record Dates: First submitted 2021-08-14; First posted 2021-08-20 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: Continuous positive airway pressure; Rho-associated coiled-coil containing kinases; Left ventricle mass
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and blood leukocyte
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Polysomography show AHI less than 15 events/h and participants do not receive any intervention include CPAP, oral appliance, or surgery for 6 months.
- OSA without CPAP group: Polysomography show AHI greater than 15 events/h and participants do not receive any intervention include CPAP, oral appliance, or surgery for 6 months.
- OSA with CPAP group: Polysomography show AHI greater than 15 events/h and participants receive CPAP more than 6 months.

SUMMARY:
The ROCK (Rho-associated coiled-coil containing kinases) play a critical role in the pathogenesis of cardiovascular diseases and left ventricle hypertrophy (LVH). ROCK activity can be used as a clinical biomarker for the diagnosis and monitoring of cardiovascular disorders. Obstructive sleep apnea (OSA) increase cardiovascular disease and LVH. Continuous positive airway pressure (CPAP) is the standard therapy for OSA. This study investigate the effect of CPAP on ROCK activity and left ventricle mass.

DETAILED DESCRIPTION:
The ROCK were discovered as downstream targets of Ras homologous A and regulate various important cellular functions, including proliferation, migration, adhesion, and apoptosis. They play a critical role in the pathogenesis of cardiovascular diseases, including cardiac fibrosis, hypertrophy, and remodeling. ROCK activity can be detected in human circulating leukocytes and could potentially be used as a clinical biomarker for the diagnosis and monitoring of cardiovascular disorders. It has been proven that higher ROCK activity is present in left ventricle hypertrophy (LVH) patients than those without LVH. Obstructive sleep apnea(OSA) is characterized by recurrent collapse of the pharyngeal airway during sleep that leads to intermittent nocturnal hypoxia, resulting in a broad range of cardiovascular morbidities, including coronary artery disease, heart failure, cardiac arrhythmias, and LVH. Continuous positive airway pressure (CPAP) is the standard therapy for OSA and several studies have shown that it can effectively reduce cardiovascular disease, but the effect of CPAP on left ventricle mass reduction is still uncertain. Previous studies demonstrated that patients with OSA had higher circulatory ROCK activity than those without OSA, but the role of CPAP on ROCK activity is not known. The circulatory leukocyte ROCK activity may be used as a clinical biomarker for cardiovascular disease and ROCK inhibitors may be used in the future as a treatment. OSA and CPAP treatment may also affect ROCK activity, the relationship between CPAP treatment, cardiac hypertrophy, and ROCK activity is important and should be clarified. Therefore, the main purpose of our study is to evaluate the effect of CPAP on ROCK activity and left ventricle mass.

ELIGIBILITY:
Inclusion Criteria:

● Subjects who complete a standard polysomnography study.

Exclusion Criteria:

* Patients who have heart failure (as determined by clinical symptoms or signs with elevated brain natriuretic peptide and echocardiography showing structural or functional abnormalities)
* Coronary artery disease (stress electrocardiography, myocardial scintigraphy, or coronary angiography proven coronary artery lesion)
* Hypertrophic cardiomyopathy
* Known infiltrative disease e.g. amyloidosis
* Chronic kidney disease severe than stage III
* Ischemic or hemorrhagic stroke
* Central sleep apnea,
* Hypoventilation syndrome (TCO2 or artery PaCO2 exceed 50 mmHg)
* Unstable hemodynamic state
* Eastern Cooperative Oncology Group Performance Status higher than grade 2
* Pregnant women will be excluded.
* Polysomnography exam showing sleep time less than 2 hours
* Patients who receive surgery or oral appliance during the study period

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who have snoring or any other symptoms of sleep breathing disorders receive a standard polysomnography study in the Chang Gung Sleep Center of Keelung.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
ROCK activity | Check baseline blood ROCK 1, ROCK 2, and MYTP-1 p/t and follow up these levels in six months later.
  Compare the change of blood ROCK 1, ROCK 2, and MYTP-1 p/t (The levels of phosphorylated to total myosin light chain phosphatase 1) among those three groups.
Left ventricle mass | Do baseline echocardiography and follow up echocardiography in six months later.
  Compare the change left ventricle mass index among those three groups.

SECONDARY OUTCOMES:
Blood pressure | Obtain initial and blood pressure six months later.
  Compare the blood pressure among those three groups.

CONTACTS AND LOCATIONS:
Overall Officials: Sleep center, Principal Investigator — Chang Gung Memorial Hospital, Keelung
Locations (1):
- Sleep center, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Requestors need application and explain the purpose. The data access will be provided after approved by review panel.

REFERENCES:
- [Background] Julian L, Olson MF. Rho-associated coiled-coil containing kinases (ROCK): structure, regulation, and functions. Small GTPases. 2014;5:e29846. doi: 10.4161/sgtp.29846. Epub 2014 Jul 10. PMID 25010901
- [Background] Sekizuka H, Osada N, Akashi YJ. Impact of obstructive sleep apnea and hypertension on left ventricular hypertrophy in Japanese patients. Hypertens Res. 2017 May;40(5):477-482. doi: 10.1038/hr.2016.170. Epub 2016 Dec 1. PMID 27904155
- [Background] Stewart MH, Lavie CJ, Shah S, Englert J, Gilliland Y, Qamruddin S, Dinshaw H, Cash M, Ventura H, Milani R. Prognostic Implications of Left Ventricular Hypertrophy. Prog Cardiovasc Dis. 2018 Nov-Dec;61(5-6):446-455. doi: 10.1016/j.pcad.2018.11.002. Epub 2018 Nov 6. PMID 30408469
- [Background] Zhang L, Zhuang JH, Peng H, Huang J, Huang LQ, Zhao ZX. Correlation between endothelial dysfunction, Rho-associated protein kinase activity, C-reactive protein and obstructive sleep apnoea syndrome in male patients. J Int Med Res. 2012;40(6):2183-90. doi: 10.1177/030006051204000616. PMID 23321175